CLINICAL TRIAL: NCT03211780
Title: Use of Intra-Operative Shear Wave Ultrasound Vibrometry for Characterization of Esophageal Malignant Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to the inability to enroll and carry out study intervention.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, MD, PhD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-002253
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: Shear wave vibrometry and B-mode imaging will be performed after esophageal distension with a fluid filled balloon intra-operatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasound (Experimental)
  Interventions: Device: General Electric LOGIQ E9 ultrasound system

INTERVENTIONS:
Device: General Electric LOGIQ E9 ultrasound system — Patients will be brought to the operating room in line with standard clinical practice and after esophageal exposure, but before surgical mobilization of the esophagus, shear wave vibrometry and B-mode imaging will be performed after esophageal distension with a fluid filled balloon intra-operatively.

SUMMARY:
Using the analysis of group velocity for a screening application and then higher order analysis based on the elastic and viscious components of the shear modulus may allow discrimination between extent of tumor invasion through the esophageal wall if appropriately correlated with pathological findings.

DETAILED DESCRIPTION:
Use of ultrasound-based vibrometry in this setting would allow for a relatively simple study and translation of clinical practice, as the same devices are already used in this setting, and operators have familiarity with the equipment. Incorporating another additional method to generate contrast for determining malignant tissue from normal based on biomechanical properties with the same probe would have benefit as an additional diagnostic modality.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Scheduled to undergo esophageal reconstruction for presumed or known esophageal cancer
* Subject is able to understand the study procedures and provide informed consent.

Exclusion Criteria:

* Subject is pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Determining malignant esophageal tissue from normal tissue | 1 week
  Determining malignant esophageal tissue from normal tissue by measurements using the General Electric LOGIQ E9 ultrasound system.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic; Matthew Urban, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials